CLINICAL TRIAL: NCT07079319
Title: Combined Effects of Muscle Energy Technique and Biofeedback Strengthening With and Without Kinesio Taping on Pain, Muscle Performance and Functional Status in Patients With Upper Crossed Syndrome
Brief Title: Effects of MET and Biofeedback Strengthening With and Without Kinesiotaping in Upper Crossed Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0165- Rabia
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
Keywords: Upper Crossed Syndrome; Biofeedback Strengthening; Kinesiotaping; Muscle Energy Technique; Muscle Performance
MeSH Terms: conditions — Neck Pain; Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET + Biofeedback Strengthening + Kinesiotaping (Experimental): Participants in this group will receive the same treatment protocol as Arm 1 (MET and biofeedback strengthening), with the addition of Kinesiotaping (KT) applied across the shoulder girdle. KT will be applied with 50-70% stretch from the anterior acromion to the opposite scapula, 3 times per week for 4 weeks. The tape will be worn for 14-16 hours per application. Standard physiotherapy (heat, ultrasound, neck isometrics, and stretching) will also be administered as part of the protocol.
  Interventions: Other: MET + Biofeedback Strengthening + Kinesiotaping
- MET + Biofeedback Strengthening (Active Comparator): Participants in this group will receive Muscle Energy Technique (MET) for the upper trapezius, levator scapulae, pectoralis major, and pectoralis minor using post-isometric relaxation technique. Additionally, they will perform biofeedback-based cranio-cervical flexion exercises using a pressure biofeedback unit (PBU). The intervention will be administered 3 times per week for 4 weeks, with a total of 12 sessions. Standard physiotherapy (heat application, ultrasound, neck isometrics, and stretching exercises) will also be provided.
  Interventions: Other: MET + Biofeedback Strengthening

INTERVENTIONS:
Other: MET + Biofeedback Strengthening + Kinesiotaping — Participants in this group will receive the same treatment protocol as Arm 1 (MET and biofeedback strengthening), with the addition of Kinesiotaping (KT) applied across the shoulder girdle. KT will be applied with 50-70% stretch from the anterior acromion to the opposite scapula, 3 times per week for 4 weeks. The tape will be worn for 14-16 hours per application. Standard physiotherapy (heat, ultrasound, neck isometrics, and stretching) will also be administered as part of the protocol.
  Arms: MET + Biofeedback Strengthening + Kinesiotaping
Other: MET + Biofeedback Strengthening — Participants in this group will receive Muscle Energy Technique (MET) for the upper trapezius, levator scapulae, pectoralis major, and pectoralis minor using post-isometric relaxation technique. Additionally, they will perform biofeedback-based cranio-cervical flexion exercises using a pressure biofeedback unit (PBU). The intervention will be administered 3 times per week for 4 weeks, with a total of 12 sessions. Standard physiotherapy (heat application, ultrasound, neck isometrics, and stretching exercises) will also be provided.
  Arms: MET + Biofeedback Strengthening

SUMMARY:
This randomised controlled trial will aim to evaluate the combined effects of Muscle Energy Technique (MET) and biofeedback strengthening, with and without Kinesiotaping (KT), on pain, posture, deep neck flexor strength, and functional status in individuals with Upper Crossed Syndrome (UCS). A total of 58 participants aged 18-40 years will be randomly allocated into two groups. Group A will receive MET and biofeedback strengthening, while Group B will receive the same intervention with the addition of KT. Treatments will be administered three times per week over a four-week period. Outcome measures will include the Numeric Pain Rating Scale (NPRS), Neck Disability Index (NDI), craniovertebral angle (CVA), rounded shoulder posture (RSP), and cranio-cervical flexion test (CCFT) using a pressure biofeedback unit. It is hypothesised that the addition of KT will result in greater improvements in pain reduction and postural correction compared to MET and biofeedback alone.

DETAILED DESCRIPTION:
This study will be a single-blinded, two-arm randomized controlled trial designed to evaluate the effects of combining Muscle Energy Technique (MET) and biofeedback-based strengthening exercises, with and without Kinesiotaping (KT), on pain intensity, postural correction, muscle performance, and functional status in individuals diagnosed with Upper Crossed Syndrome (UCS). UCS is a common postural dysfunction resulting from muscle imbalances in the upper quadrant, often associated with forward head posture, rounded shoulders, and neck pain, particularly in individuals with sedentary lifestyles.

A total of 58 participants between the ages of 18 and 40 years will be recruited through non-probability consecutive sampling from Horizon Hospital, Lahore. Participants who meet the inclusion criteria will be randomly assigned into two groups using computer-generated randomisation. Group A will receive MET and biofeedback strengthening via cranio-cervical flexion exercises. Group B will receive the same interventions with the addition of Kinesiotaping applied to the shoulder girdle. Interventions will be administered three times per week for a duration of four weeks, for a total of 12 sessions. Both groups will receive standard physiotherapy care, including heat application, therapeutic ultrasound, neck isometric exercises, and stretches for superficial neck muscles.

The primary outcomes will include pain measured by the Numeric Pain Rating Scale (NPRS), disability assessed using the Neck Disability Index (NDI), and postural parameters including craniovertebral angle (CVA) and rounded shoulder posture (RSP) assessed with a goniometer and measuring tape respectively. Deep neck flexor strength will be measured using the cranio-cervical flexion test (CCFT) with a pressure biofeedback unit (PBU).

Statistical analysis will be conducted using SPSS v25.0. The normality of the data will be assessed via the Kolmogorov-Smirnov test. Non-parametric tests (Wilcoxon signed-rank test and Mann-Whitney U test) will be used to evaluate within-group and between-group differences, respectively. The level of significance will be set at p < 0.05.

It is hypothesised that the group receiving MET and biofeedback strengthening with Kinesiotaping will demonstrate greater improvements in pain relief, postural alignment, deep neck flexor strength, and functional status compared to the group receiving MET and biofeedback strengthening alone.

This study aims to contribute to the growing evidence for multimodal physiotherapy interventions in the management of UCS and provide clinical guidance for the use of kinesiotaping as an adjunctive treatment in postural correction.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-40 years
* Both males and females
* NPRS score <7 for more than 2 months
* NDI score between 15-34
* Forward neck posture (confirmed by craniovertebral angle <48-50° measured by goniometer)
* Rounded shoulders posture (confirmed by supine lying test; if the distance between posterior aspect of acromion and plinth is >1 inch or 2.5 cm)
* Reduced deep neck flexors strength (confirmed by cranio-cervical flexion test (CCFT))

Exclusion Criteria:

* Age less than 18 or more than 40
* Recent trauma and/or hyper-flexibility
* History of cervical surgery in the last year
* History of infection (local or systemic), any dermatological condition tumor, chemotherapy, radiotherapy
* History of cervical fracture in the last year
* Radiating pain
* Positive upper limb tension tests

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale - NPRS | Baseline and 4 weeks post-intervention
  Pain intensity will be measured using the Numeric Pain Rating Scale (NPRS), a validated 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will self-report their pain levels at baseline and after 4 weeks of intervention.
Craniovertebral Angle (CVA) | Baseline and 4 weeks post-intervention
  Cervical posture will be assessed using the craniovertebral angle (CVA), measured with a universal goniometer. A greater angle indicates improved head posture. Measurements will be taken at baseline and after 4 weeks of intervention.
Rounded Shoulder Posture (RSP) Rounded Shoulder Posture (RSP) Rounded Shoulder Posture (RSP) | Baseline and 4 weeks post-intervention
  Rounded shoulder posture will be evaluated by measuring the distance from the posterior acromion to the plinth in a supine position using a measuring tape. A decrease in distance reflects improved shoulder alignment.
Deep Neck Flexor Strength (CCFT Score) | Baseline and 4 weeks post-intervention
  Deep neck flexor strength will be measured using the Craniocervical Flexion Test (CCFT) with a pressure biofeedback unit (PBU). Pressure will be increased in 2 mmHg increments from 20 mmHg to 30 mmHg. The maximum pressure level held for 10 seconds without superficial muscle compensation will be recorded.
Neck Disability Index - NDI | Baseline and 4 weeks post-intervention
  The Neck Disability Index (NDI) will be used to evaluate functional disability related to neck pain. It includes 10 sections rated 0-5, with higher scores indicating greater disability. Scores will be recorded at baseline and 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Zia, Phd Scholar, Principal Investigator — Riphah International University/ Mayo Hospital, Lahore; Rabia Afzal, MSc Student, Principal Investigator — Riphah International University
Locations (1):
- Horizon Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dr. Samarjeet Kittad DPC. Prevalence Of Upper Cross Syndrome In Students Studying For Competitive Exams Using Pressure Biofeedback. International Journal of Creative Research Thoughts (IJCRT). June 2023;11(6):g668-g78.
- [Background] Thacker D, Jameson J, Baker J, Divine J, Unfried A. Management of upper cross syndrome through the use of active release technique and prescribed exercises. Logan College of Chiropractic. 2011.
- [Background] Ashfaq R, Riaz H. Effect of Pressure biofeedback training on deep cervical flexors endurance in patients with mechanical neck pain: A randomized controlled trial. Pak J Med Sci. 2021 Mar-Apr;37(2):550-555. doi: 10.12669/pjms.37.2.2343. PMID 33679948
- [Background] Lwin NN, Myint T, Oo WM, San HH, Tun MT. EFFICACY ON PRESSURE-BIOFEEDBACK GUIDED CRANIOCERVICAL FLEXION EXERCISE IN NECK PAIN: A RANDOMIZED CONTROLLED TRIAL. Journal of Musculoskeletal Research.0(0):2150013.
- [Background] A Rayjade TY, R Chintamani, N Joshi. Comparative effectiveness of Kinesio taping and Ift in upper cross syndrome-A randomized clinical trial. Indian Journal of Forensic Medicine & Toxicology. 2020;14(3):127-32.